CLINICAL TRIAL: NCT03160989
Title: Acute and Chronic Responses to Blood Pressure After Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Larissa Aparecida Santos Matias, LARISSA APARECIDA SANTOS MATIAS - Principal Investigator, Federal University of Uberlandia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CEP UFU 002095/
Record Dates: First submitted 2017-05-03; First posted 2017-05-19 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Arterial Hypertension
Keywords: Blood pressure variability; Combined physical exercise; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postmenopausal and hypertensive women (Experimental): The intervention will consist of a single session and after ten weeks of combined physical exercises (aerobic and resisted). All volunteers will participate in the same procedure.
  Interventions: Other: physical exercises

INTERVENTIONS:
Other: physical exercises — The intervention will consist of a single session and after ten weeks of combined physical exercises (aerobic and resisted). All volunteers will participate in the same procedure.

SUMMARY:
The study will evaluate the variability of blood pressure in postmenopausal and hypertensive women after only one session and after training of ten weeks of combined physical exercises (aerobic and resisted).

DETAILED DESCRIPTION:
Before starting the training program, all the volunteers will sign the Free and Informed Consent Form (TCLE) and must present a medical certificate releasing the participation. In addition, the volunteers will respond to an anamnesis questionnaire and will undergo an anthropometric evaluation before the experimental sessions. The physical exercise program will be held three times a week for 10 weeks, containing aerobic exercise (exercise treadmill) and resistance exercises (bodybuilding). Initially, a familiarization of the ergometers used will be performed, followed by a session to evaluate the intensity of resistance exercise through a maximal repetition test (1RM), and a session to evaluate aerobic fitness through an incremental treadmill test.

Before starting the training, volunteers will perform a single exercise session, following the same exercise protocol. All the volunteers will be submitted to the evaluation of the blood pressure during 24 hours through the measurement of ambulatory blood pressure (ABPM) in three moments:

* PR: pre-training rest - the volunteers will arrive at the laboratory, will be in rest for 15 minutes and after that they will place the ABPM, without having done any exercise.
* PE: post exercise - upon arriving at the laboratory, the volunteers will be submitted to a single combined exercise session, will have a maximum interval of 20 minutes for the bath and will place the MAP device.
* CR: rest after chronic training - after the end of the 10 weeks of training, the volunteers will be submitted to ABPM, again at rest, with a maximum interval of 72 hours, between the end of the training and the placement of the device.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 50 and 70 years;
* Be in the postmenopausal phase;
* Be able to practice physical exercise on treadmill and resistance exercises (bodybuilding).
* Present stage 1 hypertension, according to the guidelines of the Brazilian Society of Hypertension
* Make use of anti-hypertensive medication, except beta-blockers
* Participants should be evaluated with a cardiologist beforehand and present a certificate attesting that they are able to perform physical activities.
* Do not present physical problems or cardiovascular complications that prevent the performance of physical exercises.

Exclusion Criteria:

* Make use of beta-blockers
* Present history of stroke or acute myocardial infarction;
* Smoking;
* Present diagnosis of Diabetes Mellitus.
* Present renal pathologies
* Use hormone replacement therapies

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in ambulatory blood pressure variability in ten weeks | After ten weeks and before ten weeks of exercise training
  The ambulatory blood pressure measurement will be performed for 24 hours. With the information obtained in this measurement, blood pressure variability will be performed.

SECONDARY OUTCOMES:
Comparison resting blood pressure | After ten weeks and before ten weeks of exercise training
  The resting blood pressure is performed after 15 minutes of sitting, measured three times and the mean is calculated for analysis
Anthropometric assessments | After ten weeks and before ten weeks of exercise training
  Body composition of the volunteers

CONTACTS AND LOCATIONS:
Overall Officials: LARISSA A SANTOS MATIAS, Graduate, Principal Investigator — Federal University of Uberlandia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gomes Anunciacao P, Doederlein Polito M. A review on post-exercise hypotension in hypertensive individuals. Arq Bras Cardiol. 2011 May;96(5):e100-109. Epub 2011 Mar 4. English, Portuguese, Spanish. PMID 21359479
- [Background] Coylewright M, Reckelhoff JF, Ouyang P. Menopause and hypertension: an age-old debate. Hypertension. 2008 Apr;51(4):952-9. doi: 10.1161/HYPERTENSIONAHA.107.105742. Epub 2008 Feb 7. No abstract available. PMID 18259027
- [Background] Puga GM, Kokubun E, Simoes HG, Nakamura FY, Campbell CS. Aerobic fitness evaluation during walking tests identifies the maximal lactate steady state. ScientificWorldJournal. 2012;2012:769431. doi: 10.1100/2012/769431. Epub 2012 May 1. PMID 22666152